CLINICAL TRIAL: NCT02240511
Title: Changes in Body Composition in Heart Failure Patients After a Resistance Exercise Program and Branched Chain Amino Acid Supplementation
Brief Title: Resistance Exercise Program and Branched Chain Amino Acid Supplementation in Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, LILIA CASTILLO MARTINEz, PhD, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CLIC003
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Heart Failure
Keywords: Body Composition; Amino Acids Supplementation; Resistance Exercise
MeSH Terms: conditions — Heart Failure | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resistance Exercise (Active Comparator): Resistance Exercise (RE) therapy was divided in four parts: stretching: arms, hands, wrists, legs, knees and ankles, each one for 10 - 20 seconds with resting intervals of 5 seconds (4 series), warming and flexion: the same muscle groups, making small circles forward and backward for 5 - 10 seconds with resting intervals of 5 seconds (4 series), resistance exercises: flexion, contractions and twisting of the same muscle groups worked in the two previous sections. In this part resistance was increased with the aid of dumbbells (500 g - 1500 g), barbells and bands, and patients performed the same exercises with 15 - 20 repetitions with resting intervals of 10 seconds. (4 series), relaxation: involved the same exercises as "stretching" to rest all muscle groups worked.
  Interventions: Other: Resistance Exercise
- RE and BCAA Supplementation (Experimental): RE: Resistance Exercise Resistance Exercise therapy was the same as in the Active Comparator
  Branched Chain Aminoacids Amino 2000 BCAA (PRONAT® laboratory) supplementation group received 180 packets of 5 grams (g)and ingested 10 g/day (5 g after breakfast and 5 g before RE)
  Interventions: Dietary Supplement: RE and BCAA Supplementation

INTERVENTIONS:
Dietary Supplement: RE and BCAA Supplementation — RE: Resistance Exercise BCAA: Branched Chain Aminoacids
  Arms: RE and BCAA Supplementation
Other: Resistance Exercise
  Arms: Resistance Exercise

SUMMARY:
Heart Failure (HF) is a complex syndrome which can include the physiological, neural hormonal and metabolic complications known as "Cardiac Cachexia" (CC). In the development of CC there is a release of catabolic cytokines (Tumor Necrosis Factor-α, interleukins 1 and 6)that cause a decrease of fat free mass and fat mass. These changes in body composition might be reversed with a therapeutic combination of resistance exercise and branched chain amino acid supplementation (BCAA). Thus the purpose of this study is evaluate changes in body composition after a resistance exercise program and BCAA supplementation in patients with HF.

DETAILED DESCRIPTION:
Heart failure (HF) is a complex syndrome which results from structural and/or functional alterations that limit the ability to respond to physiological demands(1,2).These abnormalities involve metabolic and neuro-hormonal factors such as tumor necrosis factor-α (TNF-α), one of the most important catabolic cytokines related with changes in body composition, interleukin 1 (IL-1), IL-6, interferon Y, and transmission growth factor β (3-9), which produce catabolic and anabolic imbalance and promote loss of fat free mass (FFM) with or without loss of fat mass (FM) in patients with HF. This syndrome is called "Cardiac Cachexia" (CC) (10). Signs and symptoms such as fatigue, anorexia and decreased muscle strength reflect altered body composition (9, 10). There are two possible ways to counteract these catabolic factors and restore body compartments. In one of them, protein supplementation promotes protein synthesis and inhibits proteolysis (3,11,12); in the other resistance exercise (RE) increases muscle mass and muscle strength, maintaining heart rate (13,14). Previous studies report the association of protein supplementation (15-17) and exercise (18-23) with changes in muscle strength in some cases and exercise capacity in HF patients. However, these therapies were not combined, and the studies did not provide enough information about changes in body composition. Based on these reports, our hypothesis is that the combination of RE and protein supplementation in form of branched chain amino acids (BCAA) might have an anabolic effect in patients with HF since the supplementation of BCAA could be helpful as "fuel" during the exercise and maintain the muscle mass metabolism (24).

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years
* Confirmed stable heart failure (2)

Exclusion Criteria:

* No myocardial revascularization
* Unstable angina or stroke in the previous 3 months
* With no other chronic illness which contributed to loss of muscle mass (arthritis, renal failure, cancer, HIV) previous study inclusion
* Extra cardiac conditions that made patients unable to perform exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Evaluate changes in body composition in heart failure patients after a resistance exercise program and branched chain aminoacids supplementation. | Baseline, 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Juan A Pineda, MSc, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Nestor A Sánchez, MSc, Study Director — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Lilia Castillo, PhD, Study Director — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Arturo Orea, MD, Study Director — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Rocio Cervantes, Ms, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Keirns D Candace, MD, Study Chair — Massachusetts General Hospital Interpreter Services; Carlos Ocampo, Mr, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Karla Quiroz, Ms, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Mónica Tenorio, Ms, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran; Alberto Ronquillo, Mr, Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico City, Mexico

REFERENCES:
- [Derived] Pineda-Juarez JA, Sanchez-Ortiz NA, Castillo-Martinez L, Orea-Tejeda A, Cervantes-Gaytan R, Keirns-Davis C, Perez-Ocampo C, Quiroz-Bautista K, Tenorio-Dupont M, Ronquillo-Martinez A. Changes in body composition in heart failure patients after a resistance exercise program and branched chain amino acid supplementation. Clin Nutr. 2016 Feb;35(1):41-47. doi: 10.1016/j.clnu.2015.02.004. Epub 2015 Feb 14. PMID 25726428